CLINICAL TRIAL: NCT01772537
Title: The Effect of Anesthesia on Potential Cerebrospinal Fluid (CSF) and Serum Markers of Alzheimer's Disease.
Brief Title: The Effects of Anesthesia on Patients Undergoing Surgery for Repair of a Thoracoabdominal Aneurysm.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The data did not show clear results
Sponsor: Johns Hopkins University (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: NA_00067716; 5KL2RR025006 (NIH)
Record Dates: First submitted 2013-01-17; First posted 2013-01-21 (Estimated); Results first posted 2017-02-24 (Actual); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Thoracic Aneurysm; Aneurysm Stent; Cardiopulmonary Bypass; Abdominal Aneurysm
Keywords: thoracoabdominal; aneurysm; open; stent; cardiopulmonary; abdominal; bypass
MeSH Terms: conditions — Aortic Aneurysm, Thoracic; Aortic Aneurysm, Abdominal; Aneurysm | interventions — Propofol; Isoflurane

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Open repair of thoracoabdominal aneurysms (No Intervention): These will be patients undergoing an open repair of thoracoabdominal aneurysms with or without cardiopulmonary bypass. The will be observational only.
- Stent graft repair of thoracoabdominal aneurysms isoflurane (Active Comparator): These patients are patients receiving repair of thoracoabdominal aneurysms using stent grafts. These patients will be randomized to receive isoflurane as their primary anesthetic.
  Interventions: Drug: isoflurane
- Stent graft repair of thoracoabdominal aneurysms propofol (Active Comparator): These patients are patients receiving repair of thoracoabdominal aneurysms using stent grafts. These patients will be randomized to receive propofol as their primary anesthetic.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — Intravenous anesthetic
  Arms: Stent graft repair of thoracoabdominal aneurysms propofol
Drug: isoflurane
  Arms: Stent graft repair of thoracoabdominal aneurysms isoflurane

SUMMARY:
Alzheimer's disease represents a growing public health problem in developed countries. Although the pathogenesis is not clearly defined, accumulation of extracellular amyloid, neurofibrillary tangles and neuronal loss are the hallmarks of Alzheimer's disease. The effect of anesthetic agents on changes in these proteins in humans is not well characterized, but in-vitro evidence suggests that anesthetic agents can accelerate potential pathogenic mechanisms, such as increasing amyloid formation or rates of apoptosis in cultured cells and increasing amyloid levels in mice. Human data on the effect of anesthetic agents on amyloid and tau proteins is limited to a small series of 11 patients and showed a significant increase in tau levels after exposure to anesthetics. In this study the investigators propose to measure CSF and serum biomarkers in a population of patients with normal CSF dynamics, who are undergoing surgery for repair of a thoracoabdominal aneurysm. The investigators will also obtain preliminary data on whether changes in CSF levels of these proteins are associated with postoperative delirium or cognitive change.

ELIGIBILITY:
Inclusion Criteria:

* age 21-100 years of age
* Patients presenting for surgical repair of a thoracoabdominal aneurysm
* Insertion of a CSF spinal drain for clinically indicated reason

Exclusion Criteria:

* Patients with pre-existing delirium
* Inability to speak and understand English
* Severe hearing impairment, resulting in inability to converse
* Pregnancy. Pregnancy status will be assessed using a serum pregnancy test during preoperative evaluation as part of the standard of care.

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-05; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Brown, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Stent Graft Repair Propofol: Patients have a stent graft repair receiving intravenous anesthetic - patients will be induced with 1-2mg/kg of Propofol and maintained with 25-200 mcg/kg/min of Propofol.
  Propofol: Intravenous anesthetic
- Stent Graft Repair Isoflurane: standard of care anesthetic - patients will be induced with 1-2 mg/kg of propofol and maintained with 0.5%-1.5% of isoflurane.
  isoflurane
- Open Repair: These patient will receive no intervention, just standard of care.
Period: Overall Study
Arm/Group | Stent Graft Repair Propofol | Stent Graft Repair Isoflurane | Open Repair
Started | 5 | 3 | 6
Completed | 4 | 3 | 6
Not Completed | 1 | 0 | 0
Not completed — unsuccessful lumbar drain placement | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Stent Graft Repair Propofol: Intravenous anesthetic - patients will be induced with 1-2mg/kg of Propofol and maintained with 25-200 mcg/kg/min of Propofol.
  Propofol: Intravenous anesthetic
- Open Repair: These patients received no intervention, just standard of care.
- Total: Total of all reporting groups
Arm/Group | Stent Graft Repair Propofol | Stent Graft Repair Isoflurane | Open Repair | Total
Number analyzed (Participants) | 5 | 3 | 6 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 3 | 8
  >=65 years | 2 | 1 | 3 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (13) | 62 (13) | 71 (5.3) | 65.7 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 2 | 5
  Male | 3 | 2 | 4 | 9
Region of Enrollment [Number; unit: participants]
  United States | 5 | 3 | 6 | 14

OUTCOME MEASURES:

1. Primary Outcome: Changes in Cerebrospinal Fluid (CSF) Levels of Tau
Description: Quantitative levels of tau will be measured using ELISA assay technique in pg/ml to compare the differences between the group receiving Propofol and the groups receiving Isoflurane.
  .
Time Frame: From insertion of spinal drain until removal
Population: The data for changes in CSF levels of tau are not available. The study did not have adequate funding to appropriately measure these variables.
Groups:
- Propofol: Intravenous anesthetic - patients will be induced with 1-2mg/kg of Propofol and maintained with 25-200 mcg/kg/min of Propofol.
  Propofol: Intravenous anesthetic
- Isoflurane: standard of care anesthetic - patients will be induced with 1-2 mg/kg of propofol and maintained with 0.5%-1.5% of isoflurane.
  isoflurane
Arm/Group | Propofol | Isoflurane
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Changes in CSF Levels of Amyloid
Description: Quantitative levels of amyloid will be measured using ELISA assay technique in pg/ml to compare the differences between the group receiving Propofol and the groups receiving Isoflurane.
Time Frame: From insertion of spinal drain until removal
Population: The data for changes in CSF levels of amyloid are not available. The study did not have adequate funding to appropriately measure these variables.
Arm/Group | Propofol | Isoflurane
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Participants With Delirium as Assessed by the Confusion Assessment Method (CAM)
Description: Delirium was measured using the Confusion Assessment Method and the Confusion Assessment Method- Intensive Care Unit (CAM-ICU) based upon post-operative location of patient. The patients were divided into to two groups, patients that had an open thoracoabdominal aneurysm repair versus patients that had stenting of their aneurysms. Patients that had stenting of their aneurysms were also randomized to receive either Propofol or Isoflurane as for their anesthetic.
Time Frame: Immediately after surgery and at 3 and 12 months post-op
Population: Of the 6 patients that received an open thoracoabdominal aneurysm repair 2 were found to have delirium. Of the 5 subjects that had stenting and received Propofol as their primary anesthetic, 0 were found to have delirium. Of the 3 stenting subjects that received Isoflurane as their primary anesthetic, 1 were found to have delirium.
Measure: Number; unit: participants
Groups:
- Delirum Status Post Open Thoracoabdominal Aneurysm Repair: These are participants that received open thoracoabdominal aneurysm repair instead of aneurysm stenting.
- Delerium Staus Post Stenting of Aneuryms Propofol: These are participants that received stenting of thoracoabdominal aneurysms instead of an open repair and received Propofol as their primary anesthetic.
- Stent Graft Aneurysm Repair Isoflurane: These are participants that received stenting of thoracoabdominal aneurysms instead of an open repair and received Isoflurane as their primary anesthetic.
Arm/Group | Delirum Status Post Open Thoracoabdominal Aneurysm Repair | Delerium Staus Post Stenting of Aneuryms Propofol | Stent Graft Aneurysm Repair Isoflurane
Number analyzed (Participants) | 6 | 5 | 3
participants | 2 | 0 | 1

4. Other Pre Specified Outcome: Serum Inflammatory Markers
Description: Serum inflammatory markers will be compared per anesthetic group, Propofol versus Isoflurane. A sample of 10 individuals from each group will have biomarkers measured
Time Frame: From the start of the surgery to 24 hours post-op
Population: No data is available for serum inflammatory markers. The study did not have adequate funding to appropriately measure these variables.
Arm/Group | Propofol | Isoflurane
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Groups:
- Open Thoracoabdominal Aneurysm Repair: These are patients that received open thoracabdominal aneurysm repair instead of aneurysm stenting.
Arm/Group | Stent Graft Repair Propofol | Stent Graft Repair Isoflurane | Open Thoracoabdominal Aneurysm Repair
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/3 | 0/6
Other Adverse Events (participants affected / at risk) | 0/5 | 0/3 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes